CLINICAL TRIAL: NCT05704387
Title: Restrictive- vs. Individualized Assisted Fluid Management in Patients Undergoing Major Liver Resection Surgery: A Randomized Controlled Trial
Brief Title: Restrictive- vs Individualized Goal Directed Fluid Therapy in Liver Surgery
Acronym: REVOLUTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP220682
Record Dates: First submitted 2022-07-28; First posted 2023-01-30 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2023-12

CONDITIONS: Surgery-Complications
Keywords: liver; hemodynamic optimization

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled parallel superiority trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Principal investigator, the patient, the surgeon and the outcome assessor will not know the study group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- restrictive fluid therapy group (Active Comparator): Patients in this group will have a restrictive fluid therapy (1 ml/kh/h) from anesthesia induction until end of liver resection.
  Interventions: Procedure: Restrictive fluid therapy strategy
- individualized GDFT group (Experimental): In this group, from anesthesia induction until skin closure, fluid will be given to the patients based on the recommendation of the AFM software in order to optimize patient's stroke volume (SV)
  Interventions: Procedure: individualized GDFT

INTERVENTIONS:
Procedure: individualized GDFT — In this group, from anesthesia induction until skin closure, fluid will be given to the patients based on the recommandation of the AFM software in order to optimize patient's SV
  Arms: individualized GDFT group
Procedure: Restrictive fluid therapy strategy — from anesthesia induction until end of the liver resection, patient will have a restrictive fluid therapy strategy
  Arms: restrictive fluid therapy group

SUMMARY:
"Low central venous pressure (low-CVP) or a restrictive fluid administration strategy is usually used worldwide during major liver resection surgery. Although individualized goal directed fluid therapy (GDFT) has been associated with reduced morbidity and mortality in major abdominal surgery, concerns remain on blood loss when applying GDFT in liver surgery. Indeed, GDFT could lead to a higher CVP with the risk of increased blood loss and reduced quality of the surgical field especially during liver dissection.

Since evidence is scarce, this randomized controlled trial investigates the impact of a restrictive vs an individualized GDFT strategy assisted by an assisted fluid management (AFM) system on lactate level, blood loss, and postoperative morbidity including acute kidney injury (AKI) in major liver resections."

DETAILED DESCRIPTION:
Major liver resection surgery is a frequent but complex surgery with high morbidity, even in high activity centers. The morbidity is mainly related to the size of the liver resection and to bleeding, responsible for postoperative hepatocellular failure.

Intraoperative fluid administration is a major component of the anesthetic strategy to optimize the hemodynamic status and peripheral tissue perfusion of the patient. However, high-level evidence recommendations are still lacking regarding the optimal fluid strategy in patients undergoing major liver resection.

On the one hand, it has been accepted for decades that anesthetic management should focus on minimizing intraoperative bleeding by limiting fluid administration. The objective of a ""restrictive"" fluid strategy has often been to maintain a low central venous pressure (CVP), allowing to decrease the venous pressure at the level of the suprahepatic veins and the hepatic section. The lower this pressure, the more limited the bleeding by ""backflow"". This strategy is supported by surgeons because it allows them to maintain a relatively bloodless operating field (by reducing bleeding) and thus facilitates their dissection/surgical work. Under these conditions, however, an infusion of vasopressors is often necessary to maintain adequate perfusion pressure to all organs. In addition, a ""liberal"" fluid administration is often required after liver transection to compensate for blood loss and delayed vascular filling accumulated during most of the surgical procedure. This strategy therefore potentially exposes the patient to the deleterious effects of hypovolemia as reflected by an increase in blood lactate levels. Lactate is considered an indirect marker of the degree of tissue hypoperfusion.

On the other hand, in high-risk abdominal surgery, the anesthesia community recommends a more ""individualized"" fluid strategy, based on the optimization of stroke volume also called ""goal directed fluid therapy"" (GDFT) with the aim of decreasing postoperative complications. It is now even possible to apply this strategy using a real time clinical decision support system (""assisted fluid management"" or AFM). However, the concept of GDFT assisted by AFM (GDFT-AFM) could possibly be accompanied by an increase in CVP and therefore intraoperative bleeding. However, to date, no randomized study has compared these 2 fluid therapy strategies (restrictive vs GDFT-AFM) on lactate level as the primary outcome "

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Major liver surgery

Exclusion Criteria:

-arrythmia -Linguistic barrier -Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Lactate level at the end of the surgery | Up to the end of surgenry (intraoperatively)
  lactate level measured at the end of the surgery (skin closure)

SECONDARY OUTCOMES:
Total intraoperative blood loss | Up to the end of surgenry (intraoperatively)
  We will measure blood loss at the end of the surgery
Total amount of vasopressors used during surgery | Up to the end of surgenry (intraoperatively)
  We will report the total amount of vasopressor used during surgery
Total amount of fluid used during surgery | end of the surgery
  We will report the total amount of fluid used during surgery
Incidence of acute kidney injury (AKI) | postoperative day 7
  We will report the incidence of AKI at postoperative day 7 using the KDIGO classification
Incidence of postoperative complications | postoperative day 30
  We will report the incidence of postoperative complications using the clavien dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDRE JOOSTEN, MD PhD, Principal Investigator — APHP
Locations (1):
- PAUL BROUSSE, centre hepato -biliaire, Villejuif, VAL DE MARNE, France

IPD SHARING:
Plan to Share IPD: No